CLINICAL TRIAL: NCT04570787
Title: Single-center Randomized Study Evaluating Feasibility of Routine Bladder Catheterization After Mini- Percutaneous Nephrolithotripsy (PCNL)
Brief Title: Bladder Catheterization After Mini-PCNL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04/20-н
Record Dates: First submitted 2020-08-05; First posted 2020-09-30 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Urolithiasis
Keywords: Urolithiasis; PCNL; Bladder catheterisation
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Catheterization (Active Comparator): After mini-PCNL standardized follow-up protocol supposes drainage the upper urinary tract with nephrostomy, tubeless (using ureteral stent without nephrostomy) or totally tubeless (no drainage) tactics. Bladder catheterization is not performed.
  Interventions: Procedure: Urinary bladder catheterisation
- Catheterization (Active Comparator): After mini-PCNL standardized follow-up protocol supposes drainage the upper urinary tract with nephrostomy, tubeless (using ureteral stent without nephrostomy) or totally tubeless (no drainage) tactics. The bladder is to be drained with the urethral catheter in all cases.
  Interventions: Procedure: Urinary bladder catheterisation

INTERVENTIONS:
Procedure: Urinary bladder catheterisation — Installation of Foley catheter into the urinary bladder

SUMMARY:
60 patients

Inclusion Criteria:

* age from 18 to 70 years
* Indications for mini-PCNL
* ASA score: 1-3
* Single percutaneous access to pyelocaliceal system
* Size of solitary calculus up to 2.5 cm

Exclusion Criteria:

* Active urinary tract infection
* Coagulopathy
* Clinically significant infravesical obstruction (Qmax less than 10 ml / s, PVR more than 50 ml)

DETAILED DESCRIPTION:
60 patients after PCNL will be recruited and randomized into 2 groups (30 vs 30):

* No Catheterization after mini-PCNL (study) - the bladder catheterization is not performed.
* Catheterization after mini-PCNL (control) - the bladder will be drained with the urethral catheter.

All patients will fill out the VASP in 2, 6, 12, 24 hours after mini-PCNL. Ultrasound examination of urinary bladder will be performed after mini-PCNL. All the AE will be registered.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years
* Indications for mini-PCNL
* ASA score: 1-3
* Single percutaneous access to pyelocaliceal system
* Size of solitary stone up to 2.5 cm

Exclusion Criteria:

* Active urinary tract infection
* Coagulopathy
* Clinically significant infravesical obstruction (Qmax less than 10 ml / s, PVR more than 50 ml)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
To measure the level of pain in patients | 1 day
  Filling out the VASP score after PCNL by all patients in 2, 6, 12 and 24 hours

SECONDARY OUTCOMES:
To register the AE regarding catheterization or absence of catheterization | 1 day
  Performing ultrasound examination of urinary bladder after PCNL,

CONTACTS AND LOCATIONS:
Locations (1):
- First Pavlov Saint Petersburg University, Saint Petersburg, Russia